CLINICAL TRIAL: NCT03150199
Title: A Psychological-behavioral Intervention for Physical Activity in Type 2 Diabetes
Acronym: BEHOLD-8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Associate Chief of Psychiatry for Clinical Services, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016P001597
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Results first posted 2020-03-18 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Psychology, Positive; Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Psychology + Motivational Interviewing (Experimental): Participants will complete weekly positive psychology exercises and will systematically set goals related to physical activity. Study trainers will review the positive psychology exercises on the phone each week and will use motivational interviewing techniques to facilitate goal setting.
  Interventions: Behavioral: Positive Psychology + Motivational Interviewing
- MI-Based Health Education Intervention (Active Comparator): Participants will speak on the telephone each week with a study trainer. During these calls, the trainer will provide education about a health behavior related to diabetes health (physical activity, medication adherence, diet) and will use motivational interviewing techniques to facilitate the consideration of behavior change.
  Interventions: Behavioral: MI-based Health Education Intervention

INTERVENTIONS:
Behavioral: Positive Psychology + Motivational Interviewing — Participants randomized to PP-MI will receive a treatment manual. For each session, a PP exercise will be described in the manual, with instruments and space to write about the exercise and its effects. Next, an MI section will outline specific MI-based topics (e.g., pros/cons, managing slips) and facilitate physical activity goal-setting. Following randomization, participants will engage in weekly, 30-minute phone calls over the next 8 weeks. Participants will independently complete PP exercises and MI-based goals between phone sessions and review them during phone sessions. PP and MI components will be delivered step-wise within sessions (rather than intertwined).
  Arms: Positive Psychology + Motivational Interviewing
Behavioral: MI-based Health Education Intervention — Each week, participants will learn about a different health behavior topic related to diabetes health. As an attentional control, this condition has a parallel structure to the experimental arm with a treatment manual, weekly assignments, and weekly calls to review assignments. Motivational interviewing topics (e.g., pros and cons of behavior change, importance and confidence of behavior change, identification of barriers and resources to change) will be presented related to each health behavior.
  Arms: MI-Based Health Education Intervention

SUMMARY:
The focus of this study is to examine the feasibility, acceptability, and impact of a customized, combined positive psychology and motivational interviewing (PP-MI) health behavior intervention versus a motivational interviewing (MI) health education intervention in a group of patients with type 2 diabetes (T2D).

DETAILED DESCRIPTION:
The investigators will compare a combined positive psychology and motivational interviewing (PP-MI) intervention that is adapted for patients with T2D to a motivational interviewing (MI) health education intervention. The MGH Diabetes Center and MGH primary care clinics will serve as the source of subjects for the study, with patients who have a diagnosis of T2D serving as potential participants. The investigators will enroll 60 participants, who will be randomized to either an 8-week PP-MI health behavior intervention or an 8-week MI-based health education intervention.

In this project, the investigators plan to do the following:

1. Examine the feasibility and acceptability of an 8-week, telephone-delivered health behavior intervention utilizing PP exercises and MI with systematic goal-setting.
2. Determine whether the PP-MI intervention leads to greater increases in physical activity than the MI-based education intervention in T2D patients.
3. Explore the impact of the PP-MI intervention on other psychological, behavioral, and medical outcomes, compared to the MI-based education intervention.

Participants will undergo an initial screening visit during which they will meet with study staff in person. At this visit, study eligibility will be confirmed, and eligible and willing participants will be enrolled. Following enrollment, participants will complete self-report measures, and vital signs and A1c will be measured. They then will take home and wear an accelerometer for one week, to measure baseline physical activity.

Baseline information about enrolled participants will be obtained from the patients, care providers, and the electronic medical record as required for characterization of the population. This information will include data regarding medical history (type 2 diabetes mellitus), current medical variables (conditions affecting physical activity), medications, and sociodemographic data (age, gender, race/ethnicity, living alone).

Participants will undergo a second in-person visit once adequate baseline physical activity data has been obtained. In this visit, accelerometer data will be reviewed to ensure that adequate baseline activity was captured. If so, participants will be randomized to either the PP-MI or MI-based health education intervention, then begin the study intervention. During this second in-person visit, participants will receive either a PP-MI or MI-based health education treatment manual, depending on randomization.

For the PP-MI intervention:

For each session, a PP exercise will be described in the manual, with instructions and space to write about the exercise and its effects. Next, an MI section will outline specific MI-based topics (e.g., pros/cons, managing slips) and facilitate physical activity goal-setting. At subsequent sessions, participants will review the prior week's PP exercise and learn about a new exercise, then will review the prior week's physical activity goal and set a new one.

For the MI-based health education intervention:

Each week, participants will learn about a different health behavior topic related to diabetes health. They will also be introduced to motivational interviewing topics in concert with the health behavior education topics, including medication adherence, having a heart-healthy diet, and being physically active.

Participants will complete the remaining sessions by phone approximately weekly over the next 8 weeks. Phone sessions will last approximately 30 minutes, with PP-MI and physical activity assignments completed between phone sessions. PP and MI components will be delivered step-wise within sessions (rather than intertwined) based on our experience, participant feedback, and pilot work. If a week is missed, the session will not be skipped, but rather the intervention will be completed sequentially (with participants who miss weeks then missing the final sessions), with the exception of the final call, which skips to Planning for the Future in all cases.

Participants will undergo an in-person follow-up assessment at 8 weeks. At this session, participants will repeat self-report assessments that were administered at baseline. Vital signs and a blood sample will again be collected at this in-person visit. Prior to this assessment, participants will wear an accelerometer for an additional 7 days to measure physical activity. Participants will also undergo a phone follow-up assessment at 16 weeks. During this session over the phone, participants will repeat self-report assessments that were administered at baseline. Finally, prior to this follow-up, participants will wear another accelerometer for 7 days to measure physical activity.

ELIGIBILITY:
Inclusion Criteria:

1. T2D. Eligible patients will meet American Diabetes Association (ADA) criteria for T2D (e.g., HbA1c [A1C] ≥6.5%, fasting glucose ≥126 mg/d), with diagnosis confirmed by their diabetes clinician and/or medical record review.
2. Low physical activity. Low physical activity will be defined as ≤150 minutes/week of MVPA (corresponding to ADA recommendations for moderate or greater intensity aerobic physical activity). Physical activity will be measured using a brief questionnaire adapted from the International Physical Activity Questionnaire (IPAQ).

Exclusion Criteria:

1. Cognitive impairment precluding consent or meaningful participation.
2. Lack of phone availability.
3. Inability to read/write in English.
4. Additional medical conditions (e.g., severe arthritis) that preclude physical activity.
5. Enrollment in mind-body programs, lifestyle intervention programs (e.g., cardiac rehabilitation), or other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Huffman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zambrano J, Celano CM, Chung WJ, Massey CN, Feig EH, Millstein RA, Healy BC, Wexler DJ, Park ER, Golden J, Huffman JC. Exploring the feasibility and impact of positive psychology-motivational interviewing interventions to promote positive affect and physical activity in type 2 diabetes: design and methods from the BEHOLD-8 and BEHOLD-16 clinical trials. Health Psychol Behav Med. 2020;8(1):398-422. doi: 10.1080/21642850.2020.1815538. Epub 2020 Sep 14. PMID 33763296
- [Derived] Feig EH, Harnedy LE, Celano CM, Huffman JC. Increase in Daily Steps During the Early Phase of a Physical Activity Intervention for Type 2 Diabetes as a Predictor of Intervention Outcome. Int J Behav Med. 2021 Dec;28(6):834-839. doi: 10.1007/s12529-021-09966-0. Epub 2021 Feb 11. PMID 33575971
- [Derived] Huffman JC, Golden J, Massey CN, Feig EH, Chung WJ, Millstein RA, Brown L, Gianangelo T, Healy BC, Wexler DJ, Park ER, Celano CM. A Positive Psychology-Motivational Interviewing Intervention to Promote Positive Affect and Physical Activity in Type 2 Diabetes: The BEHOLD-8 Controlled Clinical Trial. Psychosom Med. 2020 Sep;82(7):641-649. doi: 10.1097/PSY.0000000000000840. PMID 32665479

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In order to meet our goal of having 60 participants complete the intervention, we recruited 63 participants in order to account for 3 participants who were Lost to Follow-Up.
Groups:
- Positive Psychology + Motivational Interviewing: Participants will complete weekly positive psychology exercises and will systematically set goals related to physical activity. Study trainers will review the positive psychology exercises on the phone each week and will use motivational interviewing techniques to facilitate goal setting.
  Positive Psychology+Motivational Interviewing: Participants randomized to PP-MI will receive a treatment manual. For each session, a PP exercise will be described in the manual, with instruments and space to write about the exercise and its effects. Next, an MI section will outline specific MI-based topics (e.g., pros/cons, managing slips) and facilitate physical activity goal-setting. Following randomization, participants will engage in weekly, 30-minute phone calls over the next 8 weeks. Participants will independently complete PP exercises and MI-based goals between phone sessions and review them during phone sessions.
Period: Overall Study
Arm/Group | Positive Psychology + Motivational Interviewing | MI-Based Health Education Intervention
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Psychology + Motivational Interviewing | MI-Based Health Education Intervention | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (10.6) | 63.5 (9.8) | 64.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 14 | 15 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 29 | 28 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 25 | 21 | 46
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0
Physical Activity [Mean (Standard Deviation); unit: steps/day] — Measured by Actigraph accelerometer, in number of steps per day.
  steps/day | 4339 (1324) | 5025 (2446) | 4682 (1980)
Moderate-Vigorous Physical Activity [Mean (Standard Deviation); unit: minutes/day] — ActiGraph GT3X+ step counters are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness. In this trial, participants will wear the accelerometer for one week at Baseline, Week 8, and Week 16 to assess the feasibility of doing so and to ensure adequate capture of physical activity.
  minutes/day | 10.48 (9.09) | 15.21 (14.03) | 12.85 (11.96)
Sedentary Time [Mean (Standard Deviation); unit: minutes/day] — Measured by Actigraph accelerometer, in minutes per day.
  minutes/day | 524.7 (79.0) | 541.6 (100.7) | 533.2 (90.2)
Positive Affect [Mean (Standard Deviation); unit: score on a scale] — The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with medical illnesses, will be used to measure positive affect (Range: 10-50). Higher scores indicate higher levels of positive affect.
  score on a scale | 35.00 (5.74) | 37.07 (8.46) | 36.03 (7.24)
Optimism [Mean (Standard Deviation); unit: score on a scale] — Life Orientation Test-Revised is a well-validated 6-item instrument used to measure dispositional optimism (Range: 0-24). Higher scores indicate higher levels of optimism.
  score on a scale | 23.30 (4.68) | 23.27 (5.06) | 23.28 (4.83)
Self-Efficacy for Exercise [Mean (Standard Deviation); unit: score on a scale] — Measured by the Self-Efficacy for Exercise scale (SEE), a validated scale which assess self-efficacy barriers to exercise (Range: 0-90). Higher scores indicate higher efficacy expectations in relation to exercising.
  score on a scale | 54.93 (25.21) | 56.63 (17.04) | 55.78 (21.35)
Depression [Mean (Standard Deviation); unit: score on a scale] — The Hospital Anxiety and Depression Scale (HADS)-depression subscale was be used to measure depression. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Higher scores indicate higher levels of depression.
  score on a scale | 3.87 (2.99) | 3.70 (4.07) | 3.78 (3.54)
Anxiety [Mean (Standard Deviation); unit: score on a scale] — The Hospital Anxiety and Depression Scale (HADS)-anxiety subscale was be used to measure anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Higher scores indicate higher levels of anxiety.
  score on a scale | 5.53 (4.05) | 5.20 (3.72) | 5.37 (3.86)
Resilience [Mean (Standard Deviation); unit: score on a scale] — Measured by the Brief Resilience Scale (BRS), a reliable scale which assesses a person's ability to recover from stress despite adversity (Range: 6-30). Higher scores indicate more resilience.
  score on a scale | 18.00 (2.38) | 18.03 (1.83) | 18.02 (2.10)
Perceived Social Support [Mean (Standard Deviation); unit: score on a scale] — Measured by the Multidimensional Scale of Perceived Social Support (MSPSS), a scale that measures subjectively reported social support (Range: 12-84). Higher scores indicate more subjectively reported social support.
  score on a scale | 69.60 (12.46) | 69.80 (12.50) | 69.70 (12.38)
Diabetes Self-Care [Mean (Standard Deviation); unit: score on a scale] — Measured by the Summary of Diabetes Self-Care Activities (SDSCA), a well-validated measure of diabetes self-management that is associated with clinical outcomes (Range: 0-7). Higher scores indicate more diabetes self-care activities.
  score on a scale | 3.05 (1.30) | 3.02 (1.35) | 3.03 (1.31)
Medication Adherence [Mean (Standard Deviation); unit: percentage of medication taken] — Measured by Self-Reported Medication Adherence (SRMA), a two-item self-report medication adherence scale measuring percentage of time (in 10% increments) patients report taking their heart medications in the past one and two weeks. Minimum: 0, Maximum: 100. Higher scores indicate greater levels of medication adherence.
  percentage of medication taken | 90 (20) | 93 (19) | 91 (19)
Self-Reported Physical Activity [Mean (Standard Deviation); unit: MET minutes per week] — Measured by the self-report International Physical Activity Questionnaire (IPAQ). The measure assesses the types of intensity of physical activity that people do as part of their daily lives. All activities are converted to multiples of resting energy expenditure (MET) minutes per week.
  MET minutes per week | 1165.13 (2132.54) | 1017.59 (2959.11) | 1091.36 (2558.28)
Physical Function [Mean (Standard Deviation); unit: score on a scale] — Measured by the 20-item short form of the Patient-Reported Outcomes Measurement Information System (PROMIS), a well-validated measure of physical function that is highly responsive to changes in a patient's physical function status (Range: 20-100). Higher scores indicate better physical function.
  score on a scale | 92.27 (8.12) | 93.10 (7.04) | 92.68 (7.55)
Pain-Related Disability [Mean (Standard Deviation); unit: score on a scale] — Measured by the Pain Disability Index (PDI), a well-validated measure of the extent to which pain interferes with different daily activities (Range 0-70). Higher scores indicate greater interference from pain.
  score on a scale | 9.30 (10.81) | 8.73 (12.76) | 9.02 (11.73)
Weight [Mean (Standard Deviation); unit: pounds] | 196.47 (41.68) | 201.05 (41.31) | 198.76 (41.21)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.57 (6.24) | 32.38 (5.81) | 31.97 (5.99)
Blood Pressure (systolic) [Mean (Standard Deviation); unit: millimeters of mercury] | 142.7 (18.75) | 133.43 (13.48) | 138.07 (16.85)
Blood Pressure (diastolic) [Mean (Standard Deviation); unit: millimeters of mercury] | 75.73 (14.44) | 70.2 (8.05) | 72.97 (11.92)
Hemoglobin A1c [Mean (Standard Deviation); unit: mg/dL] | 7.40 (1.51) | 7.75 (1.41) | 7.57 (1.46)

OUTCOME MEASURES:

1. Primary Outcome: Number of PP-MI Sessions Completed by Participants
Description: Measured by number of PP-MI sessions completed by participants in the PP-MI group.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: sessions completed
Arm/Group | Positive Psychology + Motivational Interviewing
Number analyzed (Participants) | 30
sessions completed | 7.4 (1.8)

2. Secondary Outcome: Ease of PP Component
Description: Participants in the PP-MI group will provide ratings of ease after each PP exercise, measured on a 10-point Likert scale (0=very difficult; 10=very easy). Weekly ratings were averaged to provide an overall ease of the exercises.
Time Frame: Weeks 1-8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Psychology + Motivational Interviewing
Number analyzed (Participants) | 30
units on a scale | 8.6 (1.8)

3. Secondary Outcome: Ease of MI Component
Description: Participants in the PP-MI group will provide ratings of ease after each MI exercise, measured on a 10-point Likert scale (0=very difficult; 10=very easy). Weekly ratings were averaged to provide an overall ease of the exercises.
Time Frame: Weeks 1-8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Psychology + Motivational Interviewing
Number analyzed (Participants) | 30
units on a scale | 8.5 (1.9)

4. Secondary Outcome: Utility of PP Component
Description: Participants in the PP-MI group will provide ratings of utility after each PP exercise, measured on a 10-point Likert scale (0=not at all helpful; 10=very helpful). Weekly utility ratings were averaged to provide an overall utility score of the exercises.
Time Frame: Weeks 1-8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Psychology + Motivational Interviewing
Number analyzed (Participants) | 30
units on a scale | 8.8 (1.5)

5. Secondary Outcome: Utility of MI Component
Description: Participants in the PP-MI group will provide ratings of utility after each MI exercise, measured on a 10-point Likert scale (0=not at all helpful; 10=very helpful). Weekly utility ratings were averaged to provide an overall utility score of the exercises.
Time Frame: Weeks 1-8
Measure: Mean (Standard Deviation); unit: rating out of 10
Arm/Group | Positive Psychology + Motivational Interviewing
Number analyzed (Participants) | 30
rating out of 10 | 8.6 (2.0)

6. Secondary Outcome: Change in Moderate-Vigorous Physical Activity
Description: ActiGraph GT3X+ step counters are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness. In this trial, participants will wear the accelerometer for one week at baseline, 8 weeks, and 16 weeks to assess the feasibility of doing so and to ensure adequate capture of physical activity.
Time Frame: Change from Baseline to 8 weeks, and Baseline to 16 weeks
Population: Not all participants wore the Actigraph and provided adequate data at both follow-up time points.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 29 | 30
minutes/day
  8 weeks: number analyzed (Participants) | 28 | 28
  8 weeks | 15.72 (25.07) | 2.26 (11.86)
  16 weeks: number analyzed (Participants) | 27 | 28
  16 weeks | 10.05 (23.73) | 2.47 (8.87)

7. Secondary Outcome: Change in Physical Activity
Description: Measured by Actigraph accelerometer, in number of steps per day.
Time Frame: Change from Baseline to 8 weeks, and Baseline to 16 weeks
Population: Not all participants wore the Actigraph and provided adequate data.
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 29 | 30
steps/day
  8 weeks: number analyzed (Participants) | 28 | 28
  8 weeks | 1848 (3159) | 273 (1498)
  16 weeks: number analyzed (Participants) | 27 | 28
  16 weeks | 969 (3377) | 171 (1159)

8. Secondary Outcome: Change in Sedentary Time
Description: Measured by Actigraph accelerometer, in minutes per day.
Time Frame: Change from Baseline to 8 weeks, and Baseline to 16 weeks
Population: Not all participants wore the Actigraph and provided adequate data.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 29 | 30
minutes/day
  8 weeks: number analyzed (Participants) | 28 | 28
  8 weeks | -2.66 (66.57) | -2.95 (68.71)
  16 weeks | 2.83 (60.78) | -6.42 (68.46)

9. Secondary Outcome: Change in Positive Affect
Description: The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with medical illnesses, will be used to measure positive affect (Range: 10-50). Change was calculated by subtracting the score at baseline from the score at 8 and 16 weeks. Higher scores indicate higher levels of positive affect.
Time Frame: Change in score from Baseline to 8 weeks, and Baseline to 16 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 30 | 30
score on a scale
  8 weeks: number analyzed (Participants) | 28 | 30
  8 weeks | 3.36 (4.98) | 0.13 (5.81)
  16 weeks: number analyzed (Participants) | 30 | 28
  16 weeks | 5.80 (7.17) | 2.61 (5.88)

10. Secondary Outcome: Change in Optimism
Description: Life Orientation Test-Revised is a well-validated 6-item instrument used to measure dispositional optimism (Range: 0-24). Change was calculated by subtracting the score at baseline from the score at 8 and 16 weeks. Higher scores indicate higher levels of optimism.
Time Frame: Change in score from Baseline to 8 weeks, and Baseline to 16 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 30 | 30
score on a scale
  8 weeks: number analyzed (Participants) | 28 | 30
  8 weeks | 1.36 (2.80) | 1.00 (3.02)
  16 weeks: number analyzed (Participants) | 30 | 28
  16 weeks | 1.03 (2.57) | 1.61 (3.89)

11. Secondary Outcome: Change in Self-Efficacy for Exercise
Description: Measured by the Self-Efficacy for Exercise scale (SEE), a validated scale which assess self-efficacy barriers to exercise (Range: 0-90). Higher scores indicate higher efficacy expectations in relation to exercising. This was measured at Baseline, Week 8, and Week 16.
Time Frame: Change in score from Baseline to 8 weeks, and Baseline to 16 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 30 | 30
score on a scale
  8 weeks: number analyzed (Participants) | 28 | 30
  8 weeks | 7.18 (23.92) | -3.00 (20.13)
  16 weeks: number analyzed (Participants) | 30 | 28
  16 weeks | 6.93 (21.26) | -7.89 (19.00)

12. Secondary Outcome: Change in Depression
Description: The Hospital Anxiety and Depression Scale (HADS)-depression subscale was be used to measure depression. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Change was calculated by subtracting the score at baseline from the score at 8 and 16 weeks. Higher scores indicate higher levels of depression.
Time Frame: Change in score from Baseline to 8 weeks, and Baseline to 16 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 30 | 30
score on a scale
  8 weeks: number analyzed (Participants) | 28 | 30
  8 weeks | -0.54 (2.69) | -0.97 (2.57)
  16 weeks: number analyzed (Participants) | 30 | 28
  16 weeks | -0.83 (2.70) | -0.07 (2.69)

13. Secondary Outcome: Change in Anxiety
Description: The Hospital Anxiety and Depression Scale (HADS)-anxiety subscale was be used to measure anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Change was calculated by subtracting the score at baseline from the score at 8 and 16 weeks. Higher scores indicate higher levels of anxiety.
Time Frame: Change in score from Baseline to 8 weeks, and Baseline to 16 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | MI-Based Health Education Intervention
Number analyzed (Participants) | 30 | 30
score on a scale
  8 weeks: number analyzed (Participants) | 28 | 30
  8 weeks | -0.79 (2.08) | -0.73 (2.61)
  16 weeks: number analyzed (Participants) | 30 | 28
  16 weeks | -0.27 (2.21) | -0.57 (3.70)

14. Secondary Outcome: Change in Resilience
Description: Measured by the Brief Resilience Scale (BRS), a reliable scale which assesses a person's ability to recover from stress despite adversity (Range: 6-30). Higher scores indicate more resilience.
Time Frame: Change in score from Baseline to 8 weeks, and Baseline to 16 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 30 | 30
score on a scale
  8 weeks: number analyzed (Participants) | 28 | 30
  8 weeks | -0.43 (2.50) | -0.43 (2.10)
  16 weeks: number analyzed (Participants) | 30 | 28
  16 weeks | 0.37 (2.82) | -0.32 (2.72)

15. Secondary Outcome: Change in Perceived Social Support
Description: Measured by the Multidimensional Scale of Perceived Social Support (MSPSS), a scale that measures subjectively reported social support (Range: 12-84). Higher scores indicate more subjectively reported social support.
Time Frame: Change in score from Baseline to 8 weeks, and Baseline to 16 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 30 | 30
score on a scale
  8 weeks: number analyzed (Participants) | 28 | 30
  8 weeks | 0.68 (6.15) | -1.77 (13.57)
  16 weeks: number analyzed (Participants) | 30 | 28
  16 weeks | 3.13 (7.20) | 0.36 (9.94)

16. Secondary Outcome: Change in Diabetes Self-Care
Description: Measured by the Summary of Diabetes Self-Care Activities (SDSCA), a well-validated measure of diabetes self-management that is associated with clinical outcomes (Range: 0-7). Higher scores indicate more diabetes self-care activities.
Time Frame: Change in score from Baseline to 8 weeks, and Baseline to 16 weeks
Population: Not all participants completed all follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 30 | 30
score on a scale
  8 weeks: number analyzed (Participants) | 28 | 30
  8 weeks | 0.91 (1.00) | 0.93 (1.08)
  16 weeks: number analyzed (Participants) | 29 | 28
  16 weeks | 0.87 (1.16) | 1.11 (1.21)

17. Other Pre Specified Outcome: Change in Medication Adherence
Description: Measured by Self-Reported Medication Adherence (SRMA), a two-item self-report medication adherence scale measuring percentage of time (in 10% increments) patients report taking their heart medications in the past one and two weeks. Minimum: 0, Maximum:100. Change was calculated by subtracting the score at baseline from the score at 8 weeks and 16 weeks. Higher scores indicate greater levels of medication adherence.
Time Frame: Change in score from Baseline to 8 weeks, and Baseline to 16 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: percentage of medication taken
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 30 | 30
percentage of medication taken
  8 weeks: number analyzed (Participants) | 28 | 30
  8 weeks | 4 (16) | 0 (15)
  16 weeks: number analyzed (Participants) | 30 | 28
  16 weeks | 3 (20) | 1 (21)

18. Other Pre Specified Outcome: Change in Self-Reported Physical Activity
Description: Measured by the self-report International Physical Activity Questionnaire (IPAQ). The measure assesses the types of intensity of physical activity that people do as part of their daily lives. All activities are converted to multiples of resting energy expenditure (MET) minutes per week. Change was calculated by subtracting the score at baseline from the score at 8 and 16 weeks.
Time Frame: Change from Baseline to 8 weeks, and Baseline to 16 weeks
Population: Not all participants completed all follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: MET minutes per week
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 30 | 30
MET minutes per week
  8 weeks: number analyzed (Participants) | 28 | 30
  8 weeks | 1130.56 (2737.04) | 606.29 (4098.38)
  16 weeks: number analyzed (Participants) | 28 | 28
  16 weeks | 799.04 (2753.90) | 1090.85 (1544.04)

19. Other Pre Specified Outcome: Change in Physical Function
Description: Measured by the 20-item short form of the Patient-Reported Outcomes Measurement Information System (PROMIS), a well-validated measure of physical function that is highly responsive to changes in a patient's physical function status (Range: 20-100). Higher scores indicate better physical function.
Time Frame: Change in score from Baseline to 8 weeks, and Baseline to 16 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 30 | 30
score on a scale
  8 weeks: number analyzed (Participants) | 28 | 30
  8 weeks | 0.46 (5.30) | 2.03 (3.91)
  16 weeks: number analyzed (Participants) | 30 | 28
  16 weeks | 2.83 (5.95) | 1.93 (4.85)

20. Other Pre Specified Outcome: Change in Pain-Related Disability
Description: Measured by the Pain Disability Index (PDI), a well-validated measure of the extent to which pain interferes with different daily activities (Range 0-70). Higher scores indicate greater interference from pain.
Time Frame: Change in score from Baseline to 8 weeks, and Baseline to 16 weeks
Population: Not all participants completed follow-up questionnaires at both follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 30 | 30
score on a scale
  8 weeks: number analyzed (Participants) | 28 | 30
  8 weeks | -1.36 (12.10) | -1.27 (13.57)
  16 weeks: number analyzed (Participants) | 30 | 28
  16 weeks | -2.83 (11.47) | -1.00 (8.55)

21. Other Pre Specified Outcome: Change in Weight
Description: Measured during in-person visit at baseline and post-intervention.
Time Frame: Change from Baseline to Week 8
Population: Not all participants attended the follow-up visit at Week 8, and not all of those participants who did had their weight taken.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 25 | 28
pounds | -1.10 (4.91) | -1.43 (5.78)

22. Other Pre Specified Outcome: Change in Body Mass Index (BMI)
Description: Measured during in-person visit at baseline and post-intervention.
Time Frame: Change from Baseline to Week 8
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 25 | 28
kg/m^2 | 0.04 (0.80) | -0.27 (0.99)

23. Other Pre Specified Outcome: Change in Blood Pressure (Systolic)
Description: Measured during in-person visit at baseline and post-intervention.
Time Frame: Change from Baseline to Week 8
Population: Not all participants attended the follow-up visit at Week 8.
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 27 | 29
millimeters of mercury | -2.48 (16.20) | 0.90 (11.77)

24. Other Pre Specified Outcome: Change in Blood Pressure (Diastolic)
Description: Measured during in-person visit at baseline and post-intervention.
Time Frame: Change from Baseline to Week 8
Population: Not all participants attended the follow-up visit at Week 8.
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 27 | 29
millimeters of mercury | -1.33 (13.54) | 1.86 (6.99)

25. Other Pre Specified Outcome: Change in Hemoglobin A1c
Description: Measured during in-person visit at baseline and post-intervention.
Time Frame: Change from Baseline to Week 8
Population: Not all participants attended the follow-up visit at Week 8.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Education Intervention
Number analyzed (Participants) | 27 | 29
mg/dL | -0.21 (0.57) | -0.10 (1.25)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Adverse events are "any untoward or unfavorable medical occurrence in a human subject including any abnormal sign, symptom or disease...whether or not associated with the subject's participation in the research."
Groups:
- MI-based Health Educational Intervention: Participants will speak on the telephone each week with a study trainer. During these calls, the trainer will provide education about a health behavior related to diabetes health (physical activity, medication adherence, diet) and will use motivational interviewing techniques to facilitate the consideration of behavior change.
  MI-based Health Education Intervention: Each week, participants will learn about a different health behavior topic related to diabetes health. As an attentional control, this condition has a parallel structure to the experimental arm with a treatment manual, weekly assignments, and weekly calls to review assignments. Motivational interviewing topics (e.g., pros and cons of behavior change, importance and confidence of behavior change, identification of barriers and resources to change) will be presented related to each health behavior.
Arm/Group | Positive Psychology + Motivational Interviewing | MI-based Health Educational Intervention
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/30
Other Adverse Events (participants affected / at risk) | 5/30 | 5/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Positive Psychology + Motivational Interviewing (N=30) | MI-based Health Educational Intervention (N=30)
Unexpected chest pain (Cardiac disorders) | 1 (1) | 0 (0) — Participant was admitted to the hospital for chest pain.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Positive Psychology + Motivational Interviewing (N=30) | MI-based Health Educational Intervention (N=30)
Unexpected dizziness (General disorders) | 0 (0) | 1 (1) — Participant went to the Emergency Department (ED) for dizziness.
Unexpected chest pain (Cardiac disorders) | 1 (1) | 1 (1) — Participant went to the ED because of chest pain.
Unexpected shortness of breath and atrial fibrilation (Cardiac disorders) | 1 (1) | 0 (0) — Participant went to the ED due to unexpected shortness of breath and atrial fibrillation.
Unexpected body numbness and shoulder pain (General disorders) | 0 (0) | 1 (1) — Participant went to the ED with left-sided body numbness and shoulder pain.
Foot injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Participant reported that they injured their foot while going about their daily life activities.
Unexpected hypoglycemia (Endocrine disorders) | 2 (4) | 0 (0) — Two participants each reported two episodes of hypoglycemia. Both participants reported that they felt better after drinking orange juice.
Unexpected urethral stone (General disorders) | 1 (1) | 0 (0) — Participant went to the ED because of left plank pain due to a urethral stone.
Unexpected abdominal pain (General disorders) | 0 (0) | 1 (1) — Participant went to the ED with unexpected abdominal pain and difficulty urinating.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT03150199/Prot_SAP_000.pdf